CLINICAL TRIAL: NCT04069013
Title: Randomized Controlled Trial Comparing Surgical Outcomes Following PCNL and Mini PCNL in the Treatment of Kidney Stones
Brief Title: Standard vs Mini-PCNL for the Treatment of Stone Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of British Columbia (Other); Massachusetts General Hospital (Other); Vanderbilt University Medical Center (Other); Duke University (Other); Ohio State University (Other); Columbia University (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-589
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Urolithiasis; Kidney Stone; Kidney Calculi; Ureteral Calculi; Kidney Diseases
Keywords: Percutaneous Nephrolithotomy; PCNL
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Ureteral Calculi; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PCNL (Active Comparator): Patients receive a standard PCNL procedure using a 24 fr tract
  Interventions: Procedure: PCNL
- Mini-PCNL (Active Comparator): Patients receive a mini-PCNL procedure using a 16 fr tract
  Interventions: Procedure: PCNL

INTERVENTIONS:
Procedure: PCNL — Patients receive standard of care treatment for their urolithiasis using one of two surgical procedures, either standard PCNL or Mini-PCNL

SUMMARY:
Randomized comparison of patient outcomes following standard PCNL versus mini-PCNL.

DETAILED DESCRIPTION:
This study is a randomized controlled trial which compares the operative outcomes and complications of mini-percutaneous nephrolithotomy (mini-PCNL) versus standard PCNL for renal stones. This study will be a multi-institutional, prospective randomized controlled clinical trial with patients who have already agreed to undergo PCNL. Patients will be randomized at a 1:1 ratio to receive either standard PCNL or mini-PCNL, defined as tract sizes of 30 and 16.5 to 18 French respectively. Patients will be asked to complete pre-operative, and post-operative quality of life questionnaires, and to allow collection of one additional vial of blood for measurement of factors associated with inflammation. The participating institutions are academic medical centers in the United States and Canada that are part of the EDGE research consortium.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for PCNL at participating institutions
* Age ≥ 18 years old
* Male and female patients
* Patients of all ethnic backgrounds
* Stone size 10-20mm

Patients must be capable of giving informed consent and must be capable and willing to enroll and participate fully with the study.

Exclusion Criteria:

* Conversion to open procedure
* Multiple access tracts
* Anticoagulated or history of coagulopathy
* Preoperative ureteral stent or nephrostomy tube placement
* Technical problems/impossibility of localizing the stone on the day of intervention

Patients unable to give informed consent or unwilling to enroll or participate in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Blood loss as estimated by postoperative decreases in hemoglobin Blood loss as estimated by postoperative decreases in hemoglobin Blood Loss | Post-operative day 1
  Blood loss as estimated by postoperative decreases in hemoglobin Blood loss as estimated by postoperative decreases in hemoglobin Blood loss as estimated by postoperative decreases in hemoglobin Blood loss as estimated by postoperative decreases in hemoglobin Post-op decreases in hemoglobin

SECONDARY OUTCOMES:
Surgical outcomes | 30 Days
  Discharge time
Complication Rates | 30 Days
  Complication Rates
Renal Pelvis Pressures | Intraoperative
  Intraoperative renal pelvis pressures
Procalcitonin- Inflammatory Markers | Post operative day 1
  Procalcitonin
IL-6 Inflammatory Markers | Post operative day 1
  IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No